CLINICAL TRIAL: NCT00879879
Title: Treatment of Idiopathic Pulmonary Fibrosis With Losartan: A Pilot Project
Brief Title: Losartan in Treating Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCUSF 0108 Pilot; SCUSF-PILOT-0108 (Other: SunCoast CCOP Research Base); 5U10CA081920 (NIH)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2018-09

CONDITIONS: Precancerous Condition
Keywords: precancerous condition
MeSH Terms: conditions — Precancerous Conditions | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Losartan (Experimental): 50 mg tablets of losartan taken daily by mouth for 1 year
  Interventions: Drug: losartan

INTERVENTIONS:
Drug: losartan — 50 mg losartan taken daily by mouth in capsule form for 1 year
  Other Names: losartan potassium

SUMMARY:
RATIONALE: Losartan may be effective in treating patients with idiopathic pulmonary fibrosis.

PURPOSE: This clinical trial is studying the side effects of losartan and to see how well it works in treating patients with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the effects of losartan potassium on disease progression in patients with idiopathic pulmonary fibrosis.
* Determine the safety of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral losartan potassium daily for 1 year in the absence of disease progression or unacceptable toxicity.

Patients undergo pulmonary function tests with gas diffusion lung volumes, Carbon monoxide diffusing capacity (DLCO) tests, and 6-minute walk tests at baseline and then at 3, 6, 9, and 12 months. Patients also complete baseline/transition dyspnea index questionnaires at baseline and then at 1, 3, 6, 9, and 12 months.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age > 21 years
* Diagnosis of idiopathic pulmonary fibrosis
* Patients taking Coumadin and/or N-acetylcysteine may participate in the study
* Baseline forced vital capacity (FVC) must be greater than or equal to 50%
* Baseline 6 minute walk test distance walked must be greater than or equal to 200 meters not requiring greater than 6 lpm of oxygen

EXCLUSION CRITERIA:

* Pregnant, intending to become pregnant or breastfeeding
* Current or previous smoker of cigarettes or marijuana that recently quit within the last 6 months prior to enrollment
* Allergy or allergic reaction to Losartan or any other angiotensin II receptor blocker
* Taking losartan or any other angiotensin II receptor blocker
* Baseline systolic blood pressure < 100 mmHg
* Currently taking or has taken immunosuppressant agents within the last month such as azathioprine, cyclophosphamide, colchicine and/or prednisone
* History of lung transplant
* History of kidney failure or liver disease
* Inability to attend clinic visits

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Couluris, DO, Principal Investigator — University of South Florida
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from SunCoast Community Clinical Oncology Program (CCOP) Research Base affiliated CCOP members located in the United States.
Groups:
- Losartan: 50 mg tablets of losartan taken daily by mouth for 1 year
  losartan : 50 mg losartan taken daily by mouth in capsule form for 1 year
Period: Overall Study
Arm/Group | Losartan
Started | 20
Completed | 17
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Losartan
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 20
FVC% Predicted [Mean (Standard Deviation); unit: Percentage] | 73.96 (3.76)
DLCO% Predicted [Mean (Standard Deviation); unit: Percentage] | 43.65 (16.91)
6MWT Distance [Mean (Standard Deviation); unit: meters] | 464.89 (249.54)
Chronic O2 Supplementation [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stable or Improved Forced Vital Capacity (FVC) Response at 1 Year
Description: Forced vital capacity (FVC) must be >= 50% at baseline. Stable FVC response is defined as a -5% change in FVC from baseline up to a +5% change from baseline.
  Improved FVC response is defined as 5% or greater increase in the predicted value of FVC on pulmonary function testing following 12 months of treatment.
Time Frame: 1 year
Population: Patients who received losartan for 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan
Number analyzed (Participants) | 17
Participants
  Stable | 7
  Improved | 5
  Deteriorated | 5

2. Secondary Outcome: Number of Participants With Stable, Improved, or Deteriorated Diffusion Capacity of Carbon Monoxide (DLCO) at 1 Year
Time Frame: 1 year
Population: Patients who received losartan for 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan
Number analyzed (Participants) | 17
Participants
  Stable | 10
  Improved | 2
  Deteriorated | 5

3. Secondary Outcome: Number of Patients With Stable, Improved or Deteriorated Forced Expiratory Volume at 1 Second (%FEV1) at 1 Year
Time Frame: 1 year
Population: Patients who received losartan for 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan
Number analyzed (Participants) | 17
Participants
  Stable | 8
  Improved | 2
  Deteriorated | 7

4. Secondary Outcome: Number of Patients With Stable, Improved or Deteriorated Baseline/Transition Dyspnea Index at 1 Year
Description: This index measures a patient's degree of breathlessness related to their activities of daily living including their functional impairment and their magnitude of task and effort.
Time Frame: 1 year
Population: Patients who received losartan for 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan
Number analyzed (Participants) | 17
Participants
  Stable | 5
  Improved | 2
  Deteriorated | 10

5. Secondary Outcome: Number of Patients With Stable, Improved or Deteriorated 6-minute Walk Test Results at 1 Year
Time Frame: 1 year
Population: Patients who received losartan for 12 months.
Measure: Count of Participants; unit: Participants
Groups:
- Losartan: 50 mg tablets of losartan taken daily by mouth for 1 year
  Change in secondary markers of lung function over 12 months of losartan therapy, N=17
  N (%) Stable 6 (35.29) Improved 5 (29.41) Deteriorated 6 (-1.38)
Arm/Group | Losartan
Number analyzed (Participants) | 17
Participants
  Stable | 6
  Improved | 5
  Deteriorated | 6

ADVERSE EVENTS:
Arm/Group | Losartan
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=20)
Death due to disease progression (Immune system disorders) | 1 (1) — 1 subject died after 6 months on study. Death was deemed due to disease progression and unrelated to study procedures/study agent.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=20)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — 1 subject experienced a rash on study that resolved shortly after presentation.
Fatigue (General disorders) | 1 (1) — 1 subject experienced fatigue that resolved shortly after presentation.

LIMITATIONS AND CAVEATS:
A future phase II study is necessary to establish losartan's effect on IPF, due to a small number of patients and lack of controls to establish statistically significant efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No